CLINICAL TRIAL: NCT06302777
Title: Multifactorial Analysis of Coronary Artery Plaques Using INtracoronary IMAGing for Exploration of Atherosclerotic Determinants and Progression - the MAIN-IMAGE Registry
Brief Title: MAIN-IMAGE Registry
Acronym: MAIN-IMAGE
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Dr. med. Lena Marie Seegers, MD, Goethe University
Other Study IDs: 2023-1184
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All comers registry with patients with chronic coronary syndrome or acute coronary syndrome who underwent intracoronary imaging during cardiac catherization. The aim is to identify plaque characteristics on OCT or IVUS that are associated with adverse cardiac events including myocardial infarction and atherosclerotic progression.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing pre-intervention optical coherence tomography imaging

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS or SAP patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2028-09-26 (Estimated); Study Completion 2031-09-26 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular Events (MACE) | after 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Frankfurt University Hospital, Frankfurt am Main, Hesse
  - Frankfurt University Hospital, Frankfurt